CLINICAL TRIAL: NCT06332651
Title: Metabolic Availability of Three Protein Sources in Older and Younger Men as Measured With the Indicator Amino Acid Oxidation Method
Brief Title: Metabolic Availability in Older and Younger Men
Acronym: YOMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Responsible Party: Principal Investigator, Marco Mensink, Assistant Professor, Wageningen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NL84684.091.23
Record Dates: First submitted 2023-12-19; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Ageing
MeSH Terms: interventions — Nutritional Status; Milk

STUDY DESIGN:
Intervention Model Description: It is a parallel intervention study. The intervention does not involve a drug or biologic product, however does involve an adaptation diet and a diet with measured amino acids dissolved in water, during the test day. We investigate the amino acid metabolic availability using the IAAO method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Methionine in black beans in older men (Experimental): This group of 7 participants will have 3 test days where they consume black beans with 3 different levels of methionine and they will have 4 test days where they consume the reference amino acid mixture with 4 different levels of methionine.
  Interventions: Other: Black beans
- Methionine in black beans in younger men (Experimental): This group of 7 participants will have 3 test days where they consume black beans with 3 different levels of methionine and they will have 4 test days where they consume the reference amino acid mixture with 4 different levels of methionine.
  Interventions: Other: Black beans
- Lysine in milk or sorghum in older men (Experimental): This group of 7 participants will have 3 test days where they consume milk with 3 different levels of lysine, they will have 3 test days where they consume sorghum with 3 different levels of lysine and they will have 4 test days where they consume the reference amino acid mixture with 4 different levels of lysine.
  Interventions: Other: Milk; Other: Sorghum
- Lysine milk or sorghum in younger men (Experimental): This group of 7 participants will have 3 test days where they consume milk with 3 different levels of lysine, they will have 3 test days where they consume sorghum with 3 different levels of lysine and they will have 4 test days where they consume the reference amino acid mixture with 4 different levels of lysine.
  Interventions: Other: Milk; Other: Sorghum

INTERVENTIONS:
Other: Black beans — Black beans cooked and mashed and amino acid mixture as liquid drink to make methionine the limiting amino acid in the food consumed
  Other Names: Nutrition
  Arms: Methionine in black beans in older men; Methionine in black beans in younger men
Other: Milk — Skimmed milk as liquid drink and amino acid mixture as liquid drink to make lysine the limiting amino acid in the food consumed
  Other Names: Nutrition
  Arms: Lysine in milk or sorghum in older men; Lysine milk or sorghum in younger men
Other: Sorghum — Sorghum cooked and mashed and amino acid mixture as liquid drink to make lysine the limiting amino acid in the food consumed
  Other Names: Nutrition
  Arms: Lysine in milk or sorghum in older men; Lysine milk or sorghum in younger men

SUMMARY:
The main goal of this study is to determine the metabolic availability of methionine in black beans, lysine in sorghum and lysine in milk using the indicator amino acid oxidation method both in older and in younger men.

ELIGIBILITY:
Inclusion Criteria:

Gender: Male Age: 20-35 years or 65-80 years Body Mass Index (BMI): 18.5 - 30.0 kg/m2 Healthy as assessed with a questionnaire Regular and normal eating habits as assessed with a Food Frequency Questionnaire (FFQ) Willing to comply with study procedures and use of data Having given written informed consent

Exclusion Criteria:

Chronic disease, for example:

* Diabetes mellitus / being treated for high blood glucose
* Severe cardiovascular disease (exception: hypertension)
* Hepatic disease (e.g. hepatitis)
* Renal disease
* Cancer
* Bowel disease (e.g. inflammatory bowel disease, ulcers, bleeding)
* Pancreatitis

History of medical or surgical events that may affect GI function, and the study outcomes or disease risk for participants, for example:

* Bariatric surgery
* Gastrointestinal tract surgery
* Digestive tract disorder
* Chewing problems
* History of deep venous thrombosis without anti-coagulation medication

Medicine use that interferes with, protein metabolism, GI function and the study outcomes, for example:

* Glucose lowering drugs
* Proton pump inhibitors
* Laxatives

Habits that interfere with the study outcomes:

* Protein supplement use (current use or less than 2 weeks past use)
* Smoking
* Drug use
* Alcohol consumption >21 units/week and/or >4/day
* Following a weight-loss diet, medically prescribed diet or other diet with a low calorie intake or an unbalanced nutrient intake like a vegan or very low carbohydrate diet
* Moderate to high intense physical activity for more than 5 hours a week

Other:

* Self-reported allergy or intolerance to the tested products
* Weight loss of more than 3 kg in the 3 months prior to study screening
* Current participation in other research and <2 months prior participation in other research
* Not having a general practitioner
* Not willing to accept information-transfer concerning participation in the study , or information regarding his health to his general practitioner
* Working or doing an MSc- thesis at the department of Human Nutrition and Health at Wageningen University & Research

Ages: 20 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Metabolic availability of methionine in black beans and lysine in milk and sorghum measured with the indicator amino acid oxidation method. | 1 measurement to be calculated from repeated measurements on several test days separated by 1 week
  Indicator amino acid oxidation method is used to measure metabolic availability of the limiting amino acid by measuring the oxidation of the 13C-labelled indicator amino acid in expired breath as 13CO2 when giving different levels of the limiting amino acid. Methionine metabolic availability will be assessed in black beans and lysine metabolic availability in milk and sorghum.

CONTACTS AND LOCATIONS:
Locations (1):
- Wageningen University & Research, Wageningen, Gelderland, Netherlands